CLINICAL TRIAL: NCT06734806
Title: Evaluation of the Clinical Performance of Endocrown and Overlay Restorations: A 4-Year Retrospective Study
Brief Title: Clinical Evaluation of Endocrown and Overlay Restorations
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Haydar Albayrak, Assistant Professor, TC Erciyes University
Other Study IDs: 2024/54 12/06/2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Clinical Performance of Endodontically Treated Teeth Restored With Endocrowns and Overlays
Keywords: Endocrown; Overlay restoration; Feldspathic ceramic; CAD/CAM dentistry; Retrospective study; Clinical performance; Adhesive dentistry; Plaque index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endocrown
  Interventions: Diagnostic Test: Radiographic Imaging and Digital STL Analysis; Diagnostic Test: FDI Criteria Evaluation and Plaque Index Measurement
- Overlay
  Interventions: Diagnostic Test: Radiographic Imaging and Digital STL Analysis; Diagnostic Test: FDI Criteria Evaluation and Plaque Index Measurement

INTERVENTIONS:
Diagnostic Test: Radiographic Imaging and Digital STL Analysis — This study utilizes radiographic imaging (bitewing radiographs) and digital analysis of archived STL files to evaluate the clinical performance of endocrown and overlay restorations. The STL files are processed using Materialise 3-matic software to calculate cemented surface areas. Radiographic imaging assesses the presence of secondary caries or other failures. These diagnostic methods provide quantitative and visual data to evaluate long-term outcomes of the restorations.
Diagnostic Test: FDI Criteria Evaluation and Plaque Index Measurement — This intervention includes the evaluation of dental restorations using modified FDI criteria, assessed on a 5-point Likert scale that measures aesthetic, functional, and biological outcomes. Additionally, oral hygiene is assessed through the measurement of the plaque index, with a mean score calculated for each participant. The use of both FDI-based Likert scoring and plaque index measurements allows for a detailed evaluation of restoration performance and oral health status, combining subjective patient-reported outcomes with objective clinical metrics.

SUMMARY:
Observational Study

The goal of this observational study is to evaluate the clinical performance and patient satisfaction of endodontically treated teeth restored with endocrown and overlay restorations using feldspathic ceramic blocks over a 2 to 4-year period. The main questions this study aims to answer are:

What are the survival rates of endocrown and overlay restorations in posterior teeth after 2 to 4 years? Are there differences in biological and mechanical failure rates between endocrown and overlay restorations? How do the cemented surface areas correlate with clinical outcomes? Participants who previously received endocrown or overlay restorations will undergo a clinical evaluation, including radiographic imaging, to assess secondary caries and restoration integrity. They will also rate their satisfaction with their restorations through a standardized survey. Retrospective STL file analysis will be used to measure cemented surface areas of the restorations.

DETAILED DESCRIPTION:
This retrospective observational study aims to evaluate the clinical performance and patient satisfaction of endocrowns and overlay restorations fabricated from feldspathic ceramic CAD/CAM blocks over a period of 2 to 4 years. The study involves patients treated exclusively at the Private Ortoperio Dental Clinic in Kayseri, Turkey.

Endocrowns and overlays are widely used for restoring structurally compromised teeth. Endocrowns provide macro-retention by utilizing the pulp chamber and micro-retention through adhesive cementation, making them particularly suitable for endodontically treated teeth with limited crown height or narrow interocclusal spaces. Overlays, on the other hand, provide minimally invasive coverage while preserving the underlying tooth structure. Despite their popularity, long-term clinical data for these restorations remain limited.

The study will include 39 patients, aged between 18 and 75, who previously received endocrown or overlay restorations. Eligible participants must have functioning restorations placed at least 2 years prior, with records of digital impressions (STL files) archived at the clinic. Restorations will be evaluated using modified FDI criteria to assess aesthetic, functional, and biological outcomes. The criteria for failure include ceramic fractures, loosening, dislodgment, secondary caries, and periodontal issues. Patient satisfaction will also be measured using a Likert scale questionnaire.

Digital impressions of the cemented teeth will be analyzed using Materialise 3-matic software to calculate cemented surface areas. Additionally, the oral hygiene of participants will be assessed using the plaque index, and the mean plaque index score will be calculated for each patient. Statistical analyses will be conducted to determine potential factors affecting clinical outcomes, with methods to be determined based on data characteristics.

This study seeks to fill gaps in the literature by providing robust data on the survival rates and failure mechanisms of feldspathic ceramic endocrown and overlay restorations. Results are expected to guide clinicians in material selection and application techniques for achieving optimal outcomes in similar cases.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least one posterior tooth restored with a CEREC posterior restoration (overlay and/or endocrown) during the specified period (January 2019 to September 2022).
* The restored tooth must be functional and in normal occlusal relationship.
* Participants must have archived intraoral digital impressions (STL files) of the restored teeth.

Exclusion Criteria:

* Individuals unwilling to cooperate.
* Teeth with endocrown or overlay restorations that were extracted.
* Participants younger than 18 or older than 75 years.
* Individuals with disabilities that could impede participation.
* Participants who have moved away or are deceased.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of systemically healthy individuals aged 18 to 75 years who had at least one posterior tooth restored with a CEREC posterior restoration (endocrown and/or overlay) between January 2019 and September 2022. All restored teeth were in functional occlusion and located in a complete dental arch. Participants must have archived intraoral digital impressions (STL files) of the restored teeth. Patients were recruited from a private dental clinic specializing in restorative dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation of Restorations Using FDI Criteria | 2 to 4 years after the placement of restorations, evaluated between October 3, 2024, and October 17, 2024.
  The primary outcome measure involves scoring each restoration based on modified FDI criteria, including aesthetic, functional, and biological parameters. Two independent evaluators assessed each restoration, and a consensus score was recorded on a 5-point Likert scale.

SECONDARY OUTCOMES:
Mean Plaque Index Score for Each Participant | Assessed during clinical evaluations conducted between October 3, 2024, and October 17, 2024.
  Oral hygiene was assessed for each participant by calculating the mean plaque index score, providing an average value for oral hygiene status.
Secondary Caries Evaluation | Evaluated during clinical examinations conducted between October 3, 2024, and October 17, 2024.
  Radiographic assessment was performed to detect the presence of secondary caries under or around each restoration, and the findings were documented as part of the clinical evaluation.
Cemented Surface Area Measurement | Retrospective analysis conducted on archived STL files in November 2024.
  The cemented surface area of each restoration was calculated using STL files and analyzed with Materialise 3-matic software to correlate surface area with clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ayata M, Kucukomeroglu Oktay E, Albayrak H, Cakar M, Ozcan M. Evaluation of the clinical performance of endocrown and overlay restorations: A 4-year retrospective study. J Dent. 2025 Sep;160:105874. doi: 10.1016/j.jdent.2025.105874. Epub 2025 Jun 2. PMID 40466763